CLINICAL TRIAL: NCT01841125
Title: A 12-Week Randomized, Double-blind, Parallel-group, Placebo-controlled Trial With and Open-label, 12-week Extension, Multicenter to Evaluation of the Efficacy of Escitalopram for the Treatment of Depression in Alzheimer's Disease
Brief Title: Escitalopram for the Treatment of Depression in Alzheimer's Disease
Acronym: Escitalopram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seol-Heui Han, Clinical Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADD_E_2010
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; depressive disorder
MeSH Terms: conditions — Alzheimer Disease; Depressive Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- escitalopram (Experimental): escitalopram 15mg
  Interventions: Drug: escitalopram
- Placebo (Placebo Comparator): placebo 15mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: escitalopram — escitalopram 15mg, QD(once a day), Oral medication, 24weeks
  Other Names: lexacure Tab
  Arms: escitalopram
Drug: Placebo — placebo 15mg, QD(once a day), Oral medication
  Arms: Placebo

SUMMARY:
Purpose : to Evaluation of the Efficacy of Escitalopram for the Treatment of Depression in Alzheimer's Disease

Trial Design : A 12-week, randomized, double-blind, parallel-group, placebo-controlled trial with an open-label, 12-week extension

DETAILED DESCRIPTION:
Clinical trial agreement signed by the parties to the subjects through a process of screening. if it is consider suitable for evaluating through the selection / exclusion criteria, they will be randomly assigned to the test group or control group (placebo).

Assigned to the test group or control subjects, they will be prescribe the 5mg Escitalopram or Placebo. without regard to meals, it will be taking once a day.

and than It should be increased the capacity every two weeks by 5mg/day up to a maximum 15mg/day.

and than, on the treatment for a 8 weeks, If you don't find the side effect, Maintaining the same capacity. If you find the side effect, you should lose capacity.(10mg/day)

The test group or control subjects, will receive a doctor's examination and inspection through six visits for a 24weeks from the date of the randomly assigned participants.

ELIGIBILITY:
Inclusion Criteria:

1) over the age of 50

2) Medical diagnostic criteria must meet the standard.

1. Subject diagnosed with Alzheimer's disease in accordance with NINCDS-ADRDA Criteria.
2. Subject with three or more symptoms of the Olin depression (major depressive episode) diagnostic criteria.
3. clinical dementia rating (CDR) of 0.5 to 2
4. MMSE 10 ~ 26 (K-MMSE)
5. GDS-15 ≥ 5 points

3) When screening, Cholinesterase inhibitors taking a minimum of four weeks or more stable subject.

4) During the clinical trials, Subject does not change the capacity of Cholinesterase Inhibitors.

5) MRI or CT results within 24 months of subject with Alzheimer's disease (AD)

6) Participation in clinical trials to determine their own and written informed consent form and subject who actively perform clinical procedure including the questionnaire. But the subjects with cognitive dysfunction that cannot voluntarily make the decision, can be determined by an authorized representative to participate in.

7) Subjects must be accompanied their guardian to every visit. More than three days a week, more than 4 hours per day, spend the day with the guardian.

Exclusion Criteria:

1. If you are taking other depression drugs within 4 weeks before the start of the clinical trials(e.g. SSRI, Stablon, TCA, wellbutrin, ixel)
2. If you have any other mental illness (bipolar disorder, schizophrenia, etc.)
3. If you have a serious medical illness (heart failure, angina pectoris, myocardial infarction, arteriosclerosis, etc.) or psychiatric illness.
4. Seizures, brain surgery, organic brain disease and history of organic affective disorder and at the brain MRI, abnormalities other than brain atrophy.
5. If you have a history of the test drug hypersensitivity
6. If you are taking memantin (dementia)
7. If you participated in another clinical trial within 3 months.
8. If pregnant or fertile women, who have not received sterilization or if you do not want to use an effective method of contraception.
9. In laboratory tests, if you have kidney failure or liver failure.
10. If you have history or habitual drinking or a history of drug abuse.
11. Uncontrolled diabetes or hypertension.
12. If determined to be inappropriate for clinical trials.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in CSDD(Cornell scale for depression in dementia) from baseline after 12 weeks of between treatment groups | 12 weeks
  Change in CSDD(Cornell scale for depression in dementia) from baseline after 12 weeks of between treatment groups.

SECONDARY OUTCOMES:
Change from baseline in CSDD(Cornell scale for depression in dementia) at week 4, 8, 16 and 24. | 24weeks
  Change from baseline in CSDD(Cornell scale for depression in dementia) at week 4, 8, 16 and 24.
Change from baseline in K-MMSE at week 12 and 24. | 24 weeks
  Change from baseline in K-MMSE at week 12 and 24.
Change from baseline in ADAS-Cog at week 12 and 24. | 24 weeks
  Change from baseline in ADAS-Cog at week 12 and 24.
Change from baseline in NPIQ at week 12 and 24. | 24 weeks
  Change from baseline in NPIQ at week 12 and 24.
Change from baseline in S-IADL at week 12 and 24. | 24 weeks
  Change from baseline in S-IADL at week 12 and 24.
Change from baseline in GDS-15 at week 4, 8, 12, 16 and 24. | 24 weeks
  Change from baseline in GDS-15 at week 4, 8, 12, 16 and 24.
Change from baseline in CDR at week 12 and 24. | 24 weeks
  Change from baseline in CDR at week 12 and 24.
Change from baseline in CDR sum of box at week 12 and 24. | 24 weeks
  Change from baseline in CDR sum of box at week 12 and 24.
Change from baseline in Pittsburgh Sleep Quality Index at week 12 and 24. | 24 weeks
  Change from baseline in Pittsburgh Sleep Quality Index at week 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Seol-Heui HAN, Professor, Principal Investigator — Kunkuk Universicy Hospital; Dong-Won YANG, Professor, Principal Investigator — Seoul St. Mary's Hospital; Sung-Yoon KIM, Professor, Principal Investigator — Asan Medical Center; Kun-Woo PARK, Professor, Principal Investigator — Korea University Hospital; Do-Hoon KIM, Professor, Principal Investigator — Hanlym University Hospital; So-Young MUN, Professor, Principal Investigator — AJU University Hospital
Locations (1):
- MedicalExcellence, Seoul, Secho-gu Banpo-dong, South Korea